CLINICAL TRIAL: NCT07054008
Title: The Effect of Microsurgical Approach to Periodontal Flap Healing: A Randomized Controlled Trial
Brief Title: Microsurgery and Periodontal Healing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Angela Palaiologou-Gallis, DDS, MS, Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001809
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Periodontal Diseases
Keywords: Surgical flap treatment
MeSH Terms: conditions — Periodontal Diseases | interventions — Microsurgery

STUDY DESIGN:
Intervention Model Description: A two-arm randomized controlled split-mouth trial. Subjects will be randomized only for the first (mesial) incision to Group 1 (microscope) or Group 2 (dental loupes). The second incision (distal) will receive the other treatment. Every patient will receive both treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Microsurgical incision closure (Experimental): Microsurgical approach to wound closure using a digital microscope to enhance view
  Interventions: Procedure: Microsurgical approach with Digital Microscope
- Group 2: Dental loupes incision closure (No Intervention): Standard of care surgical approach to wound closure using Dental Loupes.

INTERVENTIONS:
Procedure: Microsurgical approach with Digital Microscope — The incision will be sutured with the use of a digital microscope (30 X) (Group 1). The microsurgical approach is a research only procedure that may add time to the total surgical time (< 6%).
  Other Names: Microsurgery
  Arms: Group 1: Microsurgical incision closure

SUMMARY:
Scientists do research to answer important questions which might help change or improve the way we do things in the future.

The investigators know that using glasses with special attachments that provide magnification (dental loupes) for dental procedures results in better healing than not using magnification. This study will test if using a microscope, that gives much higher magnification, can result in even better healing than using dental loupes.

DETAILED DESCRIPTION:
A two-arm split mouth randomized controlled trial investigating the effect of using an experimental microsurgical approach with a digital microscope (Group 1) or standard of care surgical approach with dental loupes (Group 2) on post-operative wound healing of two standardized vertical releasing incisions. The split mouth design will ensure that each patient serves as their own control.

The hypothesis is that the wound closure technique in Group 1: Microsurgical approach with digital microscope will have improved periodontal flap vertical releasing incision wound healing as compared to the Group 2: Standard of Care surgical approach with dental loupes.

ELIGIBILITY:
Inclusion Criteria:

1. Ability of subject to understand and the willingness to sign a written informed consent document.
2. Males and females; Age 18 -89 years old
3. Require surgical flap treatment of periodontal disease
4. Either maxillary or mandibular arch
5. ASA I or II
6. Has consistent transportation for all clinical and study visits

Exclusion Criteria:

1. Pregnancy, or those planning to become pregnant
2. Diabetics with an HbA1c >7.1
3. Not eligible for surgical periodontal therapy
4. Require vertical or horizontal hard tissue augmentation
5. Non-English speaking

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08-31 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Early wound healing index | One, two and three weeks
  Assessment of early soft tissue wound healing

SECONDARY OUTCOMES:
Difference in time between procedures | End of surgical procedure at last suture placement
  The time needed for suturing the incision with the digital microscope (Group 1) and with standard of care dental loupes (Group 2) will be documented immediately after placement of the last suture.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Palaiologou-Gallis, DDS, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will ensure all mechanisms used to share data will include proper plans and safeguards for the protection of privacy, confidentiality, and security for data dissemination and reuse (e.g., all data will be thoroughly de-identified and will not be traceable to a specific study participant). Plans for archiving and long-term preservation of the data will be implemented as appropriate.
Supporting Information: Study Protocol, SAP
Time Frame: At the conclusion of the study after data analysis is complete and the research is published in a peer reviewed journal